CLINICAL TRIAL: NCT06044506
Title: A Phase I Study of Autologous Natural Killer Cell Therapy for Hepatocellular Carcinoma
Brief Title: Autologous Natural Killer Cell Therapy for Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Cosphiadi Irawan, Head of Hematology-Medical Oncology Division, Dr Cipto Mangunkusumo General Hospital, Dr Cipto Mangunkusumo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22080996
Record Dates: First submitted 2023-09-01; First posted 2023-09-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Natural Killer Cell; Immunotherapy; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Autologous Natural Killer Cell (Experimental): Dosage Form: Autologous Natural Killer (NK) Cells. These cells will be harvested from the patient's body and infused back into the patient.
  Dosage: The specific dose quantity will be determined based on the patient's medical condition and response to the treatment. Customized dosages will be calculated for each individual.
  Frequency: The treatment will be given through an intravenous method.
  Duration: The length of the treatment will vary depending on how the patient responds and their medical assessment. It may take several weeks to evaluate its effectiveness and potential impacts thoroughly.
  Interventions: Drug: Autologous Natural Killer Cell Therapy; Device: Clinimacs Plus

INTERVENTIONS:
Drug: Autologous Natural Killer Cell Therapy — The therapy will be administered intravenously
Device: Clinimacs Plus — The CliniMACS Plus device is an automated cell separation tool that uses MACS Technology. It incorporates a flexible system designed for isolating clinically labeled cells using MicroBeads.

SUMMARY:
This study represents a phase I clinical trial that utilizes natural killer (NK) cell therapy for patients diagnosed with liver cancer, specifically those classified as Child-Pugh A and falling within the Barcelona Clinic Liver Cancer (BCLC) stages B or C. The expected results include determining the suitable treatment dosage, identifying any resulting side effects, and calculating the average duration of progression-free survival. The target group for the study consists of all individuals diagnosed with liver cancer. At the same time, the practical sample consists of those who received medical care for liver cancer at Cipto Mangunkusumo Hospital (RSCM) between May and December 2022. The chosen research sample comprises liver cancer patients who fulfill the predetermined participation criteria. The necessary sample size for discerning appropriate treatment dosages and the occurrence rate of potential side effects shall consist of 2-3 liver cancer patients who are administered autologous NK cells. The process for isolating these NK cells adheres to the guidelines established by Miltenyi Biotec.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-60 years old
* Patients with Hepatocellular Carcinoma (HCC) staged as BCLC B and C
* Karnofsky Performance Status (KPS) score ≥ 70
* Expected patient survival of more than three months
* The following parameters are within the normal range:

Platelet count ≥ 80,000/µL White blood cell count ≥ 3000/µL Neutrophil count ≥ 2000 Hemoglobin ≥ 9 mg/dL International Normalized Ratio (INR) 0.8-1.5 Adequate liver function (bilirubin < 2, SGOT and SGPT < 60 U/L) Adequate kidney function (serum creatinine < 1.3, serum urea < 10)

Exclusion Criteria:

* Refusing to participate in the study
* Afflicted by other malignancies, whether non-HCC liver or other malignancies
* Patients are affected by other conditions such as hypertension, severe coronary disease, myelosuppression, respiratory disorders, and acute or chronic infections
* Patients who have previously undergone transplantation and received other stem cell therapies

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Optimal treatment dosage | Start of infusion of Autologous NK cells (Day 0) until up to 6 months
  To evaluate the safety of autologous NK cell infusion and discover dose-limiting toxicities (DLT). This evaluation will determine the recommended dosage for the next trial phase.

SECONDARY OUTCOMES:
Tumor Shrinkage | Up to 6 months
  CT scans will measure tumor size at baseline and specific post-infusion times. Tumor response will be assessed using mRECIST criteria.
Immunological Responses | Up to 6 months
  Flow cytometry will evaluate infused NK cells' biomarkers, such as CD45 and CD56, that persist in peripheral blood. These biomarkers will be evaluated pre- and post-infusion.
Hematology Profile | Start of infusion of Autologous NK cells (Day 0) until up to 6 months
  Changes of Complete Blood Count (CBC), Differential Blood Count, Coagulation Profile, Mean Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amio Transferase (AST) from baseline at each assessment time point
Progression-free survival | Start of infusion of Autologous NK cells (Day 0) until progressive disease or death, whichever comes first, up to 2 years
  This metric indicates the period during which a patient's condition shows no signs of progressing or deteriorating subsequent to the administration of autologous natural killer (NK) cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: Cosphiadi Irawan, MD, PhD, Principal Investigator — Cipto Mangunkusumo Hospital/Faculty of Medicine, Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided